CLINICAL TRIAL: NCT07187453
Title: Improving Gum Health Among Older Adults in Hong Kong Through Artificial Intelligence-Based Mobile Health for Personalized Oral Hygiene Instruction
Brief Title: Improving Gum Health Among Older Adults Using AI Based mHealth for Personalized OHI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Walter Y.H. Lam, Clinical Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 25-043
Record Dates: First submitted 2025-09-18; First posted 2025-09-23 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Gum Inflammation; Periodontal Diseases; Oral Hygiene, Oral Health
Keywords: Gum Health; Oral Hygiene; Oral Health; Mobile Health; Artificial Intelligence; Elderly; Personalized Oral Hygiene Instruction
MeSH Terms: conditions — Gingivitis; Periodontal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test Group (only) (Experimental): This study is single test group (no control) study with pre vs post design. The (only) single test group will receive an intervention which involve the delivering personalized oral hygiene advice using AI assisted gum disease screening tool by non-dental personnel social workers.
  Interventions: Behavioral: Personalized Oral Hygiene Advice using AI assisted mHealth Tool by Non-Dental Personnel

INTERVENTIONS:
Behavioral: Personalized Oral Hygiene Advice using AI assisted mHealth Tool by Non-Dental Personnel — The intervention involve the delivering personalized oral hygiene advice using AI assisted gum disease screening tool by non-dental personnel social workers. Our proposed intervention involve AI to assist in the self-detection of gum disease, and emphasizes the use of mHealth for disease prevention and monitoring. Moreover, the proposed project focuses on providing personalized oral hygiene instruction, which can be utilized or provided by non-dental personnel volunteers. This combination of AI, mHealth, and personalized instruction in addition with regular service of non-dental personnel volunteers is a novel approach in managing periodontal health among older adults.

SUMMARY:
Background: Many older adults in Hong Kong lack thorough tooth cleaning and regular dental check-ups, which can lead to plaque-induced gum diseases and systemic health issues. A self-developed Mobile Health (mHealth) system, which utilizes smartphone photographs and artificial intelligence (AI), has been shown to accurately detect gum health. Personalized oral hygiene instruction (POHI) can then be provided based on the detected results.

Objectives:

1. To improve gum health among non-institutionalized older adults using mHealth and POHI.
2. To evaluate the clinical effectiveness of mHealth and POHI in improving gum health.

Hypothesis: The personalized oral hygiene instruction (OHI) in addition to AI based mHealth provided by volunteer social workers can improve clinical effectiveness and oral health related quality of life (OHRQoL).

Design and subjects: 88 older adults will be recruited from daycare centers, who will receive bi-weekly POHI based on their gum condition, detected by mHealth which is provided by trained volunteers.

Two calibrated assessors will assess the participants' gum health, oral hygiene, caries, dental plaque, and structured questionnaire at baseline, after 3 months, 6 months, 9 months and 1 year Study Instruments: Gingival Index, Plaque Index, International Caries Detection and Assessment System (ICDAS) code, dental plaque microbiology, and Geriatric Oral Health Assessment Index (GOHAI) + Structured Questionnaire.

Interventions: Personalized oral hygiene instruction using AI-powered mHealth provided by trained volunteers bi-weekly Main Outcomes: Gingival condition, Oral hygiene status, Dental plaque microbiology, and oral health-related quality of life.

Data analysis: t-tests and Wilcoxon rank-sum test will compare pre- and post-intervention data.

Expected Result: The use of mHealth and POHI provided by trained volunteers bi-weekly can lead to improved gum health among older adults.

DETAILED DESCRIPTION:
The project will be conducted in prospective design (pre- and post-) comparing before and after the intervention without sub-group. Eligible elderly will receive bi-weekly AI-based mHealth and personalized OHI provided by (non-dental) trained volunteers. The recruitment of participants among Hong Kong elderly would be according to the following pre-set criteria. The clinical effectiveness of bi-weekly AI-based mHealth and personalized OHI provided by volunteer (non dental professonial people) will be assessed by Gingival Index, Plaque Index, Dental plaque microbilology, the International Caries Detection and Assessment System (ICDAS), and Structured Questionnaire for Oral Health Related Quality of Life (OHRQoL). The time interval for intervention will be up to 1 year. The assessments will be performed at baseline and 3-month, 6-month, 9-month and 1-year intervals.

Approximately 50 volunteers will be recruited through the respective district council of the participating day care centers in Hong Kong. They will be provide a one-day training at Faculty of Dentistry, the University of Hong Kong, regarding how to operate the mHealth system, provide personalized feedback based on the AI outputs, basics of conducting the structured interviews, and communicate with the subjects.

Subjects: 88 eligible subjects will be recruited through three day-care centers in Hong Kong.

(Pre) Baseline: Written informed consent will be obtained on the day of the baseline examination. Sociodemographic information such as age, gender, education, occupation, and medical conditions will be collected. The intraoral photo of participants will be taken for reference status of baseline. Two independent assessors will assess participants' gingival health status using gingival index, oral hygiene status using plaque index and participants' caries status using ICDAS criteria. Dental plaque on surface layer of root will be carefully collected without causing pain using sterilized excavators from two sites of each participant with root caries i.e. dental plaque from the sound root surface and root caries. Each Sample will be immediately suspended in 300 μl ethanol and frozen at -80°C later until further analysis of microbiome composition. Additionally, patient's demographics and OHRQoL using structured questionnaires and Geriatric Oral Health Assessment Index (GOHAI) will be assessed.

Intervention: Participants will need to join for 3 months to 1 year. The participants will receive baseline and bi-weekly mHealth intervention to test the gum condition and receive personalized OHI to specific areas based on the result tested. Trained volunteers will take the anterior teeth and gum photo of participants with a smartphone camera at their homes or elderly centers without using any additional device such as retractors. Participants may need to pull the lips and cheek by their hands for photo taking. The photo will be uploaded into AI powered gum disease detection mobile application (GumAI app) by volunteers. The mHealth system will screen the intraoral photograph of anterior teeth, analyse the photograph, and label the gum condition as Healthy (green)/questionable (yellow)/diseased (red) within 2 minutes. According to the results tested by GumAI app, the volunteers will give personalized site specific OHI such as tooth brushing and interdental cleaning to elderly participants. This instruction includes brushing and interdental cleaning. If they have any personal concern or unclear points regarding oral hygiene practice, they can ask.

(Post) Assessment: The same assessment as in baseline at 3- months, 6 months, 9 months and 1 year will be examined by 2 calibrated dentists.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥60 years and able to give informed consent:
* Subjects who are mentally and cognitively healthy
* Subjects who have at least 20 anterior maxillary or mandibular natural teeth including incisors and canine.
* Subjects who can speak, read, or understand Cantonese for complete the satisfaction questionnaire.
* Subjects who can practice oral hygiene procedure (regular tooth brushing and interdental cleansing/flossing/brushing) daily on their own independently.

Exclusion Criteria:

* Subjects who have less than 20 anterior maxillary or mandibular natural teeth with or without dental prostheses in those area.

  * Subjects who have mental illness, or similar problems that unable to complete the satisfaction questionnaire.
  * Subjects who cannot perform oral hygiene procedure (regular tooth brushing and interdental cleansing/flossing/brushing) by any condition of oral cavity such as tumor or maxillomandibular fixation.
  * Subjects who cannot attend weekly oral hygiene instruction at centers.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Plaque Index | From enrollment (Baseline) Vs 3 months Vs 6 months Vs 9 months Vs 1 year
  Oral Hygiene status assessment using plaque index ((Silness and Loe, 1965), with a scale from 0 to 3 (higher scores mean worse outcome) on index teeth only as follow.
  0 = No plaque in the gingival area.
  1. = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface.
  2. = Moderate accumulation of soft deposits within the gingival pocket, on the gingival margin and/or adjacent tooth sur- face, which can be seen by the naked eye.
  3. = Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.
Gingival Index | From enrollment (Baseline) Vs 3months Vs 6 months Vs 9 months Vs 1 year
  Gingival health status assessment using gingival index. Dentist will perform clinical examination of anterior teeth using mouth mirror and periodontal probe to grade gingival index (gingival index (Löe H 1967), with a scale from 0 to 3, (higher scores mean worse outcome)) on index teeth.
  0 = normal gingiva;
  1. = mild inflammation: a slight change in colour, slight oedema, no bleeding on probing;
  2. = moderate inflammation: redness, oedema, glazing, or bleeding on probing;
  3. = severe inflammation: marked redness and oedema, a tendency toward spontaneous bleeding, and ulceration.

SECONDARY OUTCOMES:
Dental plaque microbiology | At baseline only (cross sectional data)
  The contents of microbiome in dental plaques from root caries will be investigated. From collected and stored plaque samples, total DNA will be extracted from pellets centrifuged using QIAamp DNA Mini Kit (Qiagen, USA). An aliquot of DNA will be used to screen the bacterial microbiome community using 16S rRNA gene V3-V4 region (~450 bp) amplicon sequencing.
International Caries Detection and Assessment System (ICDAS) for dental caries status | From enrollment (Baseline) Vs 3 months Vs 6 months Vs 9 months Vs 1 year
  (Code 0,A,B,C,E, higher scores, worse outcome) Code 0/Sound: Root surface does not exhibit any unusual discoloration that distinguishes it from the surrounding or adjacent root areas nor does it exhibit a surface defect either at the cement-enamel junction or wholly on root surface.
  Code A/Initial lesion: clearly demarcated area on the root surface or at the cement-enamel junction (CEJ) that is discolored (light/dark brown, black) but no cavitation present (loss of anatomical contour < 0.5 mm).
  Code B/Moderate lesion: clearly demarcated area on the root surface or at the CEJ that is discolored (light/dark brown, black) and cavitation (loss of anatomical contour ≥ 0.5 mm ≤ -2 mm) present.
  Code C/Extensive lesion: clearly demarcated area on the root surface or at the CEJ that is discolored (light/dark brown, black) and cavitation (loss of anatomical contour > 2mm) present.
  Code E: If for any reason a root surface cannot be visualized directly
The Geriatric Oral Health Assessment Index (GOHAI) | From enrollment (Baseline) Vs 3 months Vs 6 months Vs 9 months Vs 1 year
  A structured interview tool to evaluate participants' oral health-related quality of life. Geriatric Oral Health Assessment Index (GOHAI - Chinese Version) will be used as a structured interview tool to evaluate participants' oral health-related quality of life. 12 questionnaires focusing on patients' perspective, self-reported outcomes on behavioral, knowledge and awareness would be asked to all participants at baseline and 3- month ( using all in Chinese Version) format. The score ranges 12-60 for a 5-level scale, in which higher scores mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Lam, BDS, MDS, AdvDip Prosth, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Prince Philip Dental Hospital, Hong Kong, Central and Western District, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chau RCW, Cheng ACC, Mao K, Thu KM, Ling Z, Tew IM, Chang TH, Tan HJ, McGrath C, Lo WL, Hsung RT, Lam WYH. External Validation of an AI mHealth Tool for Gingivitis Detection among Older Adults at Daycare Centers: A Pilot Study. Int Dent J. 2025 Jun;75(3):1970-1978. doi: 10.1016/j.identj.2025.01.008. Epub 2025 Jan 26. PMID 39864975
- [Background] Chau RCW, Li GH, Tew IM, Thu KM, McGrath C, Lo WL, Ling WK, Hsung RT, Lam WYH. Accuracy of Artificial Intelligence-Based Photographic Detection of Gingivitis. Int Dent J. 2023 Oct;73(5):724-730. doi: 10.1016/j.identj.2023.03.007. Epub 2023 Apr 26. PMID 37117096
- [Background] Chau RCW, Thu KM, Chaurasia A, Hsung RTC, Lam WY. A Systematic Review of the Use of mHealth in Oral Health Education among Older Adults. Dent J (Basel). 2023 Aug 8;11(8):189. doi: 10.3390/dj11080189. PMID 37623285
- [Background] Chau RC, Thu KM, Hsung RT, McGrath C, Lam WY. Self-monitoring of Oral Health Using Smartphone Selfie Powered by Artificial Intelligence: Implications for Preventive Dentistry. Oral Health Prev Dent. 2024 Sep 23;22:327-340. doi: 10.3290/j.ohpd.b5758200. PMID 39308412